CLINICAL TRIAL: NCT03924531
Title: Promoting Adherence to Anti-Hypertensive Medications and Lifestyle Guidelines Through Mindfulness Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-000411
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2019-04

CONDITIONS: Health Behavior Modification Using Mindfulness
Keywords: Hypertension; Health Behavior; Mindfulness; Meditation
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Awareness Program (Experimental): The group that received mindfulness training.
  Interventions: Behavioral: Mindful Awareness Program
- Health Promotion Program (Active Comparator): The group that received the health information.
  Interventions: Behavioral: Health Promotion Program

INTERVENTIONS:
Behavioral: Mindful Awareness Program — 2-hour mindfulness training for 6 weeks.
  Other Names: Mindfulness training
  Arms: Mindful Awareness Program
Behavioral: Health Promotion Program — Health Promotion Program
  Arms: Health Promotion Program

SUMMARY:
Adherence is a major problem for the approximately one-third of Americans over the age of 20 who suffer from Hypertension (HTN). Hypertension can be controlled through medication adherence and lifestyle modifications (diet and exercise). However, nearly 50% of those with HTN report poor adherence to their antihypertensive medications, lifestyle changes, or both as primary reasons for failing to control their blood pressure. Currently, behavioral interventions are limited to providing education or reminding individuals to take better care of themselves by starting and adhering to proper diet and exercise program. Given the lack of adherence reported, education and reminders alone may not be sufficient to promote health behavior change. Interventions that appeal to individual's internal drive may be more effective, given that behavior adoption and maintenance are usually associated with intrinsic motivation and volition. Mindfulness practice is an intervention that shows promise in changing lifestyle behaviors. The purpose of this study is to investigate the use of UCLA's Mindful Awareness Program (UCLAMAP) on promoting self-management behaviors, specifically adherence to medication, diet, and exercise for those individuals with HTN. We will randomize 52 individuals with HTN who have difficulty with adherence to antihypertensive medications and lifestyle changes to the intervention group or the attention-control group. The intervention includes six sessions of the mindfulness training through UCLA's Mindful Awareness Research Center (MARC).

ELIGIBILITY:
Inclusion Criteria:

* over 21 years of age
* able to understand and speak English
* self-report of having difficulty with a healthy diet and engaging in regular physical activity.

Exclusion Criteria:

* On chemotherapy for cancer treatment
* Current substance abuse disorder (i.e., drugs, alcohol).
* Current diagnoses of Post-traumatic stress disorders, severe anxiety, or severe depression.
* On hemodialysis.
* Pregnant. (Pregnant women may develop Preeclampsia, which is a pregnancy complication characterized by high blood pressure)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Diet | up to 12 weeks
  21 item questionnaire called Rapid Eating and Activity Assessment for Patients (REAP). Various questions related to food choices. The answer choices were rarely, sometimes, and often for each food questions.
Exercise | up to 12 weeks
  The instrument used was called the Brief Physical Assessment. The is a 6 item weekly questionnaire that asked the minutes the participants performed a particular exercise behavior.
Blood pressure medication adherence | up to 12 weeks
  The instrument used was called the Brief Medication Questionnaire (BMQ).The tool includes a 5-item Regimen Screen that asks patients how they took each medication in the past week, a 2-item Belief Screen that asks about drug effects and bothersome features, and a 2-item Recall Screen about potential difficulties remembering. We collected the number of missed medication days.

SECONDARY OUTCOMES:
Blood pressure measurements | up to 12 weeks
  The participants were provided with blood pressure monitors to take home and log their blood pressure measurements daily. Blood pressure measurements were collected weekly. Systolic and diastolic blood pressure measurements will be accessed.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No